CLINICAL TRIAL: NCT06614283
Title: Effectiveness of Advance Health Mobile APP for the Self Management of Diabetes Type2 in a Resource-constrained Setting, a Randomized Control Trial
Brief Title: Advance Health Mobile APP for the Self Management of Diabetes Type2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Putra Malaysia (Other)
Responsible Party: Principal Investigator, Arshed Muhammad, PhD, Universiti Putra Malaysia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: BMU
Record Dates: First submitted 2024-09-23; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Two-arm randomized control trial
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators are blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention arm (Experimental): Ae mobile application tailored for patients with Type 2 diabetes, aiming to enhance their self-management practices will be used for the intervention arm. The app includes features such as medication tracking, appointment scheduling, patient data storage, advice for treatment and follow-ups, health education and promotion, and real-time health monitoring.
  Interventions: Behavioral: Diabetes self management @ click
- Control arm (No Intervention): The control arm will be given no intervention except usual care

INTERVENTIONS:
Behavioral: Diabetes self management @ click — A mobile application tailored for patients with Type 2 diabetes, aiming to enhance their self-management practices will be used for the intervention arm. The app includes features such as medication tracking, appointment scheduling, patient data storage, advice for treatment and follow-ups, health education and promotion, and real-time health monitoring.
  Arms: Intervention arm

SUMMARY:
Digital health using mobile health (mHealth) tools, such as telehealth and text messaging, and or mobile Apps can improve blood glucose levels in patients with type 2 diabetes. This intervention is designed to improve self-management of diabetes and blood glucose levels in diabetic patients.

DETAILED DESCRIPTION:
Patients with type 2 diabetes may experience improvements in their blood glucose levels thanks to mHealth technologies like mobile apps and telehealth text messaging. The goal of this intervention is to help diabetic people better control their blood glucose levels and diabetes. The intervention arm will employ a smartphone application designed specifically for individuals with Type 2 diabetes, with the goal of improving their self-management behaviors. Features of the app include real-time health monitoring, appointment scheduling, medication tracking, patient data storage, treatment and follow-up recommendations, and health education and promotion.

ELIGIBILITY:
Inclusion Criteria:

* The presence of T2D and at least 1 recorded HbA1c level of 8.0% or higher in the past 6 months
* Age between ages 21 and 85 years,
* Receiving primary care at the clinical site
* Having fluency in English/ Urdu in reading and writing
* Having a smartphone
* Agreeing to take part in the study

Exclusion Criteria:

* Planning to move away from the study site
* Being pregnant or in lactation, (6) being unable to send or read text messages on a mobile phone,
* Having a history of receiving or planning surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1600 (Estimated)
Dates: Start 2024-10-05 (Estimated); Primary Completion 2025-05-15 (Estimated); Study Completion 2025-06-10 (Estimated)

PRIMARY OUTCOMES:
Diabetes Self-Management | 6- months from baseline
  DSMQ-R will assess Diabetes self-management. The DSMQ-R is a multidimensional questionnaire with 27 items regarding essential self-management practices for T1D and T2D (including diabetes-adjusted eating, glucose testing/monitoring, medication taking, physical activity, and cooperation with the diabetes team). 4 Subscales:
  * 'Glucose Management' (GM), 11 items: 1, 4, 6, 10, 12, 21, 22, 23, 24, 26, 27 (10 and 12 must be inverted).
  * 'Dietary Control' (DC), 7 items: 2, 5, 9, 13, 17, 18, 25 (5, 13 and 18 must be inverted).
  * 'Physical Activity' (PA), 3 items: 8, 11, 15 (11 and 15 must be inverted).
  * 'Health-Care Use' (HU), 4 items: 3, 7, 14, 19 (7 and 14 must be inverted). SCALE SCORE = ACTUAL SUM OF ITEMS / MAXIMUM POSSIBLE SUM OF ITEMS x 10

SECONDARY OUTCOMES:
Hemoglobin A1C | 6- months from baseline
  Hemoglobin A1C will be measured by taking blood samples.
Adherence to medication | 6- months from baseline
  SEAMS URDU VERSION WILL BE USED FOR SEAMS Urdu version. It is of 13 questions with a score ranging from 13-39. Higher scores show better adherence
Health related quality of life | 6- months from baseline
  Health-related quality of life will be assessed by EQ 5D3L. The EQ-5D-3L Index score summarizes each possible health state on a numerical scale ranging from -0.594 to 1, where a score of 1 indicates full health and scores of 0 and less than 0 indicate a state equivalent to being dead, and a state

CONTACTS AND LOCATIONS:
Locations (1):
- Said Mitha Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No
Only study protocol, statistical plan, and results will be shared by publications in peer reviewed journals

REFERENCES:
- [Background] Nelson LA, Greevy RA, Spieker A, Wallston KA, Elasy TA, Kripalani S, Gentry C, Bergner EM, LeStourgeon LM, Williamson SE, Mayberry LS. Effects of a Tailored Text Messaging Intervention Among Diverse Adults With Type 2 Diabetes: Evidence From the 15-Month REACH Randomized Controlled Trial. Diabetes Care. 2021 Jan;44(1):26-34. doi: 10.2337/dc20-0961. Epub 2020 Nov 5. PMID 33154039
- [Background] Saydah S, Cowie C, Eberhardt MS, De Rekeneire N, Narayan KM. Race and ethnic differences in glycemic control among adults with diagnosed diabetes in the United States. Ethn Dis. 2007 Summer;17(3):529-35. PMID 17985509
- [Background] Choudhry NK, Isaac T, Lauffenburger JC, Gopalakrishnan C, Lee M, Vachon A, Iliadis TL, Hollands W, Elman S, Kraft JM, Naseem S, Doheny S, Lee J, Barberio J, Patel L, Khan NF, Gagne JJ, Jackevicius CA, Fischer MA, Solomon DH, Sequist TD. Effect of a Remotely Delivered Tailored Multicomponent Approach to Enhance Medication Taking for Patients With Hyperlipidemia, Hypertension, and Diabetes: The STIC2IT Cluster Randomized Clinical Trial. JAMA Intern Med. 2018 Sep 1;178(9):1182-1189. doi: 10.1001/jamainternmed.2018.3189. PMID 30083727
- [Background] American College of Clinical Pharmacy; McBane SE, Dopp AL, Abe A, Benavides S, Chester EA, Dixon DL, Dunn M, Johnson MD, Nigro SJ, Rothrock-Christian T, Schwartz AH, Thrasher K, Walker S. Collaborative drug therapy management and comprehensive medication management-2015. Pharmacotherapy. 2015 Apr;35(4):e39-50. doi: 10.1002/phar.1563. PMID 25884536